CLINICAL TRIAL: NCT05012449
Title: Transitional Ankle Fracture Management Using a New Joystick Technique
Acronym: Transitional
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Fuzhou No 2 Hospital (Other)
Responsible Party: Principal Investigator, Shunyou Chen, Clinical Professor, The Fuzhou No 2 Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Shunyou
Record Dates: First submitted 2021-07-30; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-07

CONDITIONS: Tibial Fracture
Keywords: Arthrography, Joystick technique, Adolescent, Ankle fracture
MeSH Terms: conditions — Tibial Fractures; Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthrography-assisted joystick technology. (Experimental): Adolescent transitional ankle fracture who were treated with the arthrography-assisted joystick technology.
  Interventions: Procedure: Arthrography-assisted joystick technology.
- No arthrography-assisted joystick technology. (No Intervention): Adolescent transitional ankle fracture who were treated with open or close reduction .

INTERVENTIONS:
Procedure: Arthrography-assisted joystick technology. — Arthrography-assisted joystick technology.
  Other Names: No arthrography-assisted joystick technology.
  Arms: Arthrography-assisted joystick technology.

SUMMARY:
To investigate the feasibility and short-term clinical efficacy of the arthrography-assisted joystick technique for the treatment of adolescent transitional ankle fracture.

DETAILED DESCRIPTION:
Adolescent transitional ankle fracture who were treated with the arthrography-assisted joystick technology.

ELIGIBILITY:
Inclusion Criteria:

1. X-ray or computed tomography (CT) diagnosis of adolescent transitional ankle fracture.
2. After manual reduction, the displacement of both ends of the epiphyseal plate or articular surface fracture in any direction was still > 2 mm; the arthrography-assisted joystick technique was used for treatment.

Exclusion Criteria:

1. Bilateral fracture.
2. In association with epiphyseal dysplasia and neuromuscular disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic union | Through study completion, an average of 0.5 year.
  The time of radiographic union

SECONDARY OUTCOMES:
American Orthopedic Foot and Ankle Society (AOFAS) ankle score system. | Through study completion, an average of 0.5 year.
  The AOFAS evaluation criteria were used to evaluate ankle function and healing: 90-100 points = an excellent outcome; 75-89 points = a good outcome; 50-74 points = a fair outcome; and < 50 points = a poor outcome. The scoring criteria include pain, functional and autonomic activity, support, maximum walking distance, ground walking, abnormal gait, forefoot activity, hindfoot activity, ankle-hindfoot stability, and foot alignment.

OTHER OUTCOMES:
Measurement methods of the mechanical axis of lower limbs . | Through study completion, an average of 0.5 year.
  Quantitative indicators included the full length of the tibia, the angle formed by the mechanical axis of the lower limbs in standing position and the horizontal line, and the angle of ankle mortise in coronal and sagittal positions.

CONTACTS AND LOCATIONS:
Overall Officials: Shunyou Chen, doctor, Study Chair — The Fuzhou No 2 Hospital
Locations (1):
- Shunyou Chen, Fuzhou, Fujian, China